CLINICAL TRIAL: NCT04811274
Title: Study of Macrophage Function and of the GM-CSF Signaling Pathway in Alveolar Proteinosis by Mutations of the MARS Gene
Brief Title: Macrophages, GM-CSF and MARS Proteinosis
Acronym: MacroMARS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201476; 2020-A02750-39 (Other: IDRCB number)
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Alveolar Proteinosis (PAP); MARS; Genetic Mutation
Keywords: Pulmonary alveolar proteinosis (PAP); Mutations in the MARS gene; Methionyl-tRNA synthetase; Surfactant clearance; Alveolar macrophages
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Bronchoalveolar lavage fluid (BALF)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Minor patients with alveolar proteinosis by mutations of the MARS gene.
  Interventions: Biological: Blood collection; Biological: Bronchoalveolar lavage fluid collection
- Controls: Minors patients without alveolar proteinosis.
  Interventions: Biological: Blood collection; Biological: Bronchoalveolar lavage fluid collection

INTERVENTIONS:
Biological: Blood collection — 2 to 5 ml
Biological: Bronchoalveolar lavage fluid collection — 5 to 25 ml

SUMMARY:
Mutations in the MARS gene encoding methionyl-tRNA synthetase are responsible for a genetic form of alveolar proteinosis (PAP), but the pathophysiological mechanisms of the respiratory phenotype are not known.

The main hypothesis is that the PAP phenotype in these patients is secondary to a defective clearance of the surfactant by the alveolar macrophages.

The main objective of the study is to study the clearance capacity of lipoproteinaceous material by macrophages of patients with MARS related PAP. This will be investigate in cultured macrophages derived from peripheral blood monocytes of patients (patients with MARS related PAP) and controls (patients without MARS related PAP).

DETAILED DESCRIPTION:
Pulmonary alveolar proteinosis (PAP) is a rare respiratory disease characterized by the accumulation of lipoproteinaceous material within the pulmonary alveoli, resulting in the majority of cases from a defective clearance of the surfactant by intra-alveolar macrophages.

Mutations in the MARS gene encoding methionyl-tRNA synthetase are responsible for a genetic form of alveolar proteinosis, but the pathophysiological mechanisms leading to mutations in the respiratory phenotype are not known.

The main hypothesis is that the alveolar proteinosis phenotype in these patients is secondary to a defective clearance of the surfactant by the alveolar macrophages.

The main objective of the study is to study the clearance capacity of lipoproteinaceous material by macrophages of patients with MARS related PAP. This will be investigate in cultured macrophages derived from peripheral blood monocytes of patients (patients with MARS related PAP) and controls (patients without MARS related PAP).

The subjects and the controls will be included during a hospitalization during which a blood sample and a bronchoscopy with broncoalveolar lavage must be performed as part of their care.

ELIGIBILITY:
Inclusion Criteria:

* Minors from 0 to 17 years hospitalized for their care at Necker Enfants Malades hospital and for whom a blood sample and a bronchoscopy with bronchoalveolar lavage must be performed as part of their care
* Information and consent of the holders of parental authority and the patient

Exclusion Criteria:

- Refusal of holders of parental authority or patient

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor patients with alveolar proteinosis by mutations of the MARS gene and minor patients without alveolar proteinosis, hospitalized for their care at Necker Enfants Malades hospital and for whom a blood sample and a bronchoscopy with bronchoalveolar lavage must be performed for their care.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2021-11-06 (Actual)

PRIMARY OUTCOMES:
Measurement of the clearance | Day 0
  Measurement of the clearance of abnormal lipo-proteinaceous material (from patients) at 48h of culture by cultured macrophages derived from peripheral blood monocytes from patients and controls.
  Microscopic examination of cell samples prepared on slide after cytospin and stained with oil red'O.

SECONDARY OUTCOMES:
Measurement of the clearance after supplementation with methionine | Day 0
  Measurement of the clearance of abnormal lipo-proteinaceous material (from patients) at 48h culture with methionine supplementation in culture medium by cultured macrophages derived from peripheral blood monocytes from patients and controls.
  Microscopic examination of cell samples prepared on slide after cytospin and stained with oil red'O.
Cellular phenotyping and study of the GM-CSF pathway | Day 0
  Description : Study the impact of mutations on the cell phenotype and the GM-CSF signalling pathway.
  (i) CD11b and CD49d cell immunostaining which are surface markers of healthy alveolar macrophages ; (ii) measurement of the level of intracellular phosphorylation of STAT5 by flow cytometry; and (iii) measurement of the level of expression of the SPI1, PPARγ and ABCG1 genes by quantitative PCR.
  These measurements will be performed in cultured macrophages derived from peripheral blood monocytes of patients and controls, but also in alveolar macrophages directly isolated from the BAL fluid of patients and controls. All these measurements will be performed in response to incubation with GM-CSF.

CONTACTS AND LOCATIONS:
Overall Officials: Alice HADCHOUEL, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No